CLINICAL TRIAL: NCT07297901
Title: Headache Calm: App-based Breathing Program for Migraine Relief
Brief Title: App-based Breathing Program for Migraine Relief
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Sunny Wonsun Kim, Ph.D, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00023014
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Migraine; Heart Rate Variability (HRV); Autonomic Nervous System; Headache (Migraine); Headache; Chronic Pain; mHealth; Breathing
Keywords: heart rate variability biofeedback; migraine; headache; chronic pain; remotely delivered
MeSH Terms: conditions — Migraine Disorders; Headache; Chronic Pain; Respiratory Aspiration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline and HRVB (Experimental): Participants will complete an online baseline survey and 28 days of baseline daily headache diary assessments prior to random assignment to the HRVB arm. This group will receive a standardized HeartMath© Inner Balance device by mail. Participants will attend a 30-40-minute one-on-one HRVB training session via Zoom prior to initiating the HRVB intervention and will be asked to practice HRV biofeedback at home for 10 minutes per day over an eight-week period.
  Participants will receive an email or phone notification as a weekly reminder to complete their at-home HRVB practice. At the end of the 8-week intervention period, participants will be scheduled for a follow-up Zoom meeting to collect a 5-minute post-intervention resting HRV measurement and will complete the T2 online survey.
  Interventions: Behavioral: Baseline Survey; Behavioral: Heart rate variability biofeedback
- Baseline and Sham Control Group (Sham Comparator): Participants will complete an online baseline survey and 28 days of baseline daily headache diary assessments prior to randomization to the sham control arm. Participants will receive a standardized HeartMath© Inner Balance device by mail and will attend a 30-40-minute one-on-one sham training session via Zoom before initiating the sham intervention. They will be instructed to engage in normal breathing at home for 10 minutes per day over an eight-week period, without receiving HRV biofeedback or real-time visualization. Weekly email or phone reminders will be provided to support adherence. At the end of the 8-week intervention period, participants will attend a follow-up Zoom visit to complete a 5-minute post-intervention resting HRV measurement and the T2 online survey.
  Interventions: Behavioral: Baseline Survey; Behavioral: Sham Control Group

INTERVENTIONS:
Behavioral: Baseline Survey — Baseline surveys contain a series of scaled questions, including sociodemographic variables (age, sex, etc), information about migraine frequency and intensity, Insomnia Severity Index (ISI), Grade Chronic Pain Scale Revised (GCPS-R), Pain Catastrophizing Scale (PCS), Emotional Regulation Questionnaire (ERQ), Depression Anxiety Stress Scale-21 (DASS-21), and treatment expectations.
Behavioral: Heart rate variability biofeedback — Participants randomized to the intervention arm will receive a standardized HRV sensor and accompanying smartphone application, along with a 30-40-minute HRVB training session focused on using biofeedback signals to generate a resonant frequency pattern of HRV (coherence) following baseline data collection. Participants will be asked to practice their HRVB skills at home for 10 minutes per day over a 8-week period.
  Arms: Baseline and HRVB
Behavioral: Sham Control Group — Participants randomized to the sham control arm will receive a standardized HRV sensor and accompanying smartphone application, along with a 30-40-minute sham breathing training session following baseline data collection. Participants will be asked to practice their sham breathing exercises at home for 10 minutes per day over an 8-week period.
  Arms: Baseline and Sham Control Group

SUMMARY:
Migraine is one of the most common neurological disorders, characterized by recurrent headaches, sensitivity to light and movement, nausea, and autonomic dysregulation. Although mind-body interventions like biofeedback have shown their efficacy, they remain underutilized due to barriers such as transportation, time constraints, lack of awareness, stigma, and cost. A targeted approach to enhancing HRV is HRV biofeedback (HRVB), a technique using visual or auditory feedback to help people regulate HRV through slow-paced breathing and positive emotional regulation to promote ANS balance and emotional resilience. Investigators will conduct a remotely delivered pilot RCT of an 8-week, 10 min/day, novel app-based HRVB intervention compared to a sham control intervention (matching intervention time and attention with no biofeedback component) in adult with chronic migraine. Investigators hypothesize data collected from the study will: a) support the feasibility and acceptability of the remotely delivered app-based HRVB intervention among adults with chronic migraine, and b) provide insights into refining the intervention by examining patterns of change in migraine and psychological outcomes from pre- to post-intervention.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aimed at examining the effect of Heart Rate Variability Biofeedback (HRVB) among people with chronic migraine. The primary objective of the study is to determine whether HRVB can positively impact the psychosocial health and well-being of those living with chronic migraines. Building upon our prior pilot RCT (IRB study ID: STUDY00018977; ClinicalTrials.gov ID: NCT06546163), which demonstrated the feasibility and acceptability of HRVB in college-aged women with disordered eating, investigators propose to examine the feasibility of a HRVB intervention using the device investigators have successfully implemented remotely, incorporating video guides and Zoom-based coaching for smartphone app set-up and use. Investigators will conduct a remotely delivered pilot RCT of an 8-week, 10 min/day, novel app-based HRVB intervention compared to a sham control intervention (matching intervention time and attention with no biofeedback component) in adult with chronic migraines. There will be 30 participants who experience chronic migraines that will participate in the study and they will be randomly assigned to either the HRVB intervention group or the control group (15 for each group). Participants will first attend a baseline orientation meeting during which they complete baseline measures and will be asked to complete 28 days of a 5-10 minute daily diary survey about their migraine-related experiences. After the 28 days, participants will attend a zoom training meeting during which they complete a 5-minute heart rate measurement using a small earlobe sensor device that investigators will mail to participants , will be randomly assigned to the HRVB group or sham control group, and be asked to complete the daily diary assessments for another 28 days. After 8 weeks since the baseline and 4 weeks since group assignment, participants will attend a final zoom meeting to complete follow-up measures and the heart rate measurement. Investigators hypothesize data collected from the study will: a) support the feasibility and acceptability of the remotely delivered app-based HRVB intervention among adults with chronic migraines, and b) provide insights into refining the intervention by examining patterns of change in migraine and psychological outcomes from pre- to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 years or older
2. Chronic migraine as determined by the Identify Chronic Migraine (ID-CM) assessment
3. Access to a smartphone and Wi-Fi
4. Fluent in English.

Exclusion Criteria:

1. Major medical (e.g., cancer, HIV/AIDS) or psychiatric illness (e.g., schizophrenia)
2. Conditions that would potentially interfere with accurate detection of HRV data (i.e., medications that alter heart rhythms, indications of cardiac conduction abnormalities [e.g., heart arrhythmias], having a pacemaker or heart transplant)
3. Any form of mind-body intervention (3 or more times per week) during the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Migraine Frequency at 28 days | One month after baseline (T2), 8 weeks after baseline (4 weeks after T2) (T3)
  Migraine frequency will be assessed by the change from baseline in monthly (28-day) migraine days or moderate/severe headache days, assessed by the end of day headache daily diary .

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | Baseline (T1) and 8 weeks after baseline (T3)
  An individual's pain experience will be measured using the Pain Catastrophizing Scale (PCS) (13 items, 5-point Likert scale; 0=not at all, 4= all the time ). The PCS has three subscales: rumination, magnification, and helplessness. The PCS has been used and validated in studies of psychosocial interventions for migraine patients. Individual scores on the PCS can range from 0 to 52 with higher scores indicating a worse pain experience . (Cronbach's a = .87).
Emotional Regulation Questionnaire | Basline (T1) and 8 weeks after baseline (T3)
  Emotional regulation strategies will be measured using the Pain Catastrophizing Scale (ERQ) (10 items, 7-point Likert scale; 1= strongly disagree, 7= strongly agree). The ERQ has two subscales: cognitive reappraisal and expressive suppression. The ERQ has been used and validated in studies of psychosocial interventions for migraine patients. Individual scores on the PCS can range from 10 to 70 with higher scores indicating a greater frequency of use of emotional regulation strategies (Cronbach's a = 0.76-0.83).
Changes from 1-month after baseline (T2) Heart Rate Variability measurement at T3 | One month after baseline (T2), 8 weeks after baseline (4 weeks after T2) (T3)
  The InnerBalance from HeartMath will be used to collect HRV data using a 5-minutes "neutral" protocol (we call "waiting at the bus stop" implying that no particular intent for breath or mindful state is to be evoked) to understand the benefits of HRVB. In addition, HRV measures will be obtained for the 10-minute paced breathing period per day to understand the effects of paced breathing on migraine during the intervention period. The following precautions will be provided as instructions to participants prior to data collection: no coffee, tea, or caffeinated drinks such as energizing drinks in the 2 hours before the data collection, and no alcohol consumption during 24 hours prior to the data collection.
Depression Anxiety Stress Scale - Short Form (DASS-21) | Baseline (T1) and 8 weeks after baseline (T3)
  General psychological distress will be measured using the Depression Anxiety Stress Scale (DASS-21) (21 items, 4-point Likert scale; 0= Did not apply to me at all, 3= Applied to me very much). The ERQ has three subscales: depression, anxiety, and stress. The ERQ has been used and validated in studies of psychosocial interventions for migraine patients. Individual scores on the DASS-21 can range from 0 to 63 with higher scores indicating greater levels of general psychological distress (Cronbach's a = 0.74).
Insomnia Severity Index (ISI) | Baseline (T1) and 8 weeks after baseline (T3)
  Severity of insomnia will be measured using the Insomnia Severity Index (ISI) (7 items, 5-point Likert scale; 0=None, 4=Very severe). The ISI has been used and validated in studies of psychosocial interventions for migraine patients. Individual scores on the DASS-21 can range from 0 to 28 with higher scores indicating more sever insomnia (Cronbach's a = 0.74).
Graded Chronic Pain Scale-Revised (GCPS-R) | Baseline (T1) and 8 weeks after baseline (T3)
  Chronic pain severity will be measured using the Graded Chronic Pain Scale-Revised (GCPS-R) (5 items, 5-point Likert scale; 0 = Not at all, 4 = Extremely). The GCPS-R is one of the most frequently used and validated scales in studies of psychosocial interventions for migraine patients.The scores on the GCPS-R can can be classfied form Grade 0 (no chronic pain) to Grade 3 (high impact chronic pain) (Cronbach's a = 0.87-0.94).

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States